CLINICAL TRIAL: NCT04928651
Title: Clonidine for Analgesia to Preterm Infants During Neonatal Intensive Care - a Prospective Pharmacokinetic/Pharmacodynamic/Pharmacogenetic Observational Study. Cohort 2 in The SANNI Project
Brief Title: Clonidine for Analgesia to Preterm Infants During Neonatal Intensive Care
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Karolinska Institutet (Other); Helsinki University Central Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Örebro University, Sweden (Other); The Swedish Research Council (Other Government); University of Tartu (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-005091-26
Record Dates: First submitted 2018-03-23; First posted 2021-06-16 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-02

CONDITIONS: Intensive Care, Neonatal; Analgesia; Hypnotics and Sedatives
MeSH Terms: conditions — Agnosia | interventions — Clonidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clonidine: Preterm infants (< gw 37+0) who are in need for analgesic or sedative medication will receive treatment with clonidine according to an algorithm based on pain and sedative scoring results
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — Clonidine will be administered to preterm infants in need of analgesia and sedation; either as the primary drug for comfort and light sedation or as an "add-on" drug to opioids according to an algorithm based on pain and sedative scoring results. Opioids are mostly given to postoperative patients. These drugs (morphine or fentanyl) will not be studied, but a baseline PK sample will be taken to correlate to the baseline aEEG.

SUMMARY:
A prospective pharmacokinetic (PK), pharmacodynamic (PD) and pharmacogenetic (PG) observation study, including the PK/PD/PG relationship, in clonidine administered for analgesia and sedation to preterm newborn infants receiving neonatal intensive care. Phase 3 - therapeutic confirmatory study

DETAILED DESCRIPTION:
All preterm infants that are admitted to the study neonatal intensive care units (NICUs) for neonatal intensive care are potential study patients, and their parents will be asked for consent.

The patient will be treated according to clinical guidelines and will be included in the study if in need for clonidine according to clinical judgment (pain scores) and as decided by the responsible clinical doctor. The dosing and administration of the drug will be implemented according to an algorithm based on pain scoring results.

Apart from extra blood sampling, the bedside monitoring, investigations (electroencephalography, EEG, echocardiography, ECG, ultrasound of the brain) and follow-up (neurologic examination and magnetic resonance imaging, MRI) are the same as for all preterm infants according to local and national guidelines.

In total 100 infants will be included.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (< gw 37+0) who are in need for analgesic or sedative medication according to clinical judgment (scoring with pain assessment scales; ALPS-Neo and Comfort-Neo)
* Existing arterial or venous cannulas/catheters for repeated non-traumatic blood sampling
* Informed and written parental consent

Exclusion Criteria:

* Hemodynamic instability (same as in clinical routine).
* Cardiac malformations in need for postnatal surgery.
* Any serious medical condition or ethical issues that could, in the Investigators opinion, interfere with the study procedures.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sick preterm infants admitted to the NICU in need for analgesic or sedative medication according to clinical judgment.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of clonidine; S-concentration | Repeated blood samples (5 minutes after the loading dose, just before start of the clonidine infusion and at 1 hour, 24 hours, 48 hours and 72 hours after start of the infusion
  Clonidine analyses will be performed with LC-MS standard assay on a Waters ultra-pressure liquid chromatography (UPLC)-MS/MS system and then statistically analysed with NONMEM (Non-linear Mixed Effect Modelling) populationbased PK statistics
Pharmacokinetics (PK) of clonidine; elimination half-time | Data from repeated blood samples (5 minutes after the loading dose, just before start of the clonidine infusion and at 1 hour, 24 hours, 48 hours and 72 hours after start of the infusion
  Statistical analyses will be performed with NONMEM (Non-linear Mixed Effect Modelling) populationbased PK statistics
Pharmacokinetics (PK) of clonidine; clearance | Data from repeated blood samples (5 minutes after the loading dose, just before start of the clonidine infusion and at 1 hour, 24 hours, 48 hours and 72 hours after start of the infusion
  Statistical analyses will be performed with NONMEM (Non-linear Mixed Effect Modelling) populationbased PK statistics
Pharmacokinetics (PK) of clonidine; volume of distribution | Data from repeated blood samples (5 minutes after the loading dose, just before start of the clonidine infusion and at 1 hour, 24 hours, 48 hours and 72 hours after start of the infusion
  Statistical analyses will be performed with NONMEM (Non-linear Mixed Effect Modelling) populationbased PK statistics
Neurophysiologic amplitude-integrated EEG response in relation to PK | From 30 minutes before start of treatment until 72 hours after start of treatment.
  Analyse of single cortical events and their dynamics, based on burst detection and measuring features of individual bursts as well as their mass statistical behaviour over time.
Neurophysiologic amplitude-integrated EEG response; longer term brain function in relation to PK | From 30 minutes before start of treatment until 72 hours after start of treatment.
  Assessment of longer term brain function using measures of long range correlation and brain activity cycling.
Neurophysiologic amplitude-integrated EEG response; assessment of global brain network function in relation to PK | From 30 minutes before start of treatment until 72 hours after start of treatment.
  Assessment of global brain network function will be based on Activation Synchrony Index.

SECONDARY OUTCOMES:
Change in/association between heart rate in relation to PK . | From 30 minutes before start of treatment until 72 hours.
  The heart rate will be monitored 1/second according to clinical routine in the neonatal intensive care, and concomitantly downloaded into the aEEG (amplitude integrated electroencephalography) monitor. The change will be described as percentage increase/decrease
Change in/association between blood pressure (systolic, diastolic and mean arterial blood pressure) in relation to PK . | From 30 minutes before start of treatment until 72 hours.
  The blood pressure will be monitored 1/second according to clinical routine in the neonatal intensive care, and concomitantly downloaded into the aEEG (amplitude integrated electroencephalography) monitor. The change will be described as percentage increase/decrease
Change in/association between peripheral oxygen saturation in relation to PK . | From 30 minutes before start of treatment until 72 hours.
  The peripheral oxygenation will be monitored 1/second according to clinical routine in the neonatal intensive care, and concomitantly downloaded into the aEEG (amplitude integrated electroencephalography) monitor. The change will be described as percentage increase/decrease
Change in NIRS (near-infrared spectroscopy) response in relation to PK . | From 30 minutes before start of treatment until 72 hours.
  The NIRS registration will be sampled into a USB and downloaded and analysed. The change will be described as percentage increase/decrease
Change in pain, stress and behavioral state as assessed with a pain scale for continuous pain/stress (Astrid Lindgrens and Lund childrens hospitals Pain and stress assessment scale for Preterm and Sick newborn infants, ALPS-Neo) in relation to PK. | From 30 minutes before start of treatment until 72 hours.
  Change in pain responses as measured by pain assessment scores for continuous pain/stress, The Astrid Lindgren and Lund Children's Hospitals Pain and Stress Assessment Scale for Preterm and sick Newborn Infants (ALPS-Neo) in relation to PK. This scale evaluates facial expression, breathing pattern, tone of extremities, hand/foot activity and level of activity, rated 0-2. Will be assessed hourly according to clinical routine. The relation to PK will be analysed with the help of NONMEM statistics
Change in pain, stress and behavioral state as assessed with a pain scale for continuous pain/stress (The COMFORT-Neo scale) in relation to PK | From 30 minutes before start of treatment until 72 hours.
  Change in pain responses as measured by pain assessment scores for continuous pain/stress, the Comfort Neo, in relation to PK. This scale evaluates alertness, calmness/agitation, respiratory response, crying, body movement, facial tension and muscle tone, rated 0-5. Will be assessed hourly according to clinical routine. The relation to PK will be analysed with the help of NONMEM statistics
Procedural pain response in relation to PK: assessed with change in galvanic skin response | At one occasion during the study period (72 hours) when the analgesic treatment has not been changed the last six hours.
  Procedural pain response at a short standardized pain stimulation; as assessed with change in galvanic skin response in relation to PK. The change will be described as percentage increase/decrease
Procedural pain response in relation to PK: change in serum-cortisol | At one occasion during the study period (72 hours) when the analgesic treatment has not been changed the last six hours.
  Procedural pain response at a short standardized pain stimulation; change in serum-cortisol in relation to PK. The relation to PK will be analysed with NONMEM statistics.
Procedural pain response in relation to PK as assessed with the Premature Infant Pain Profile - revised, PIPP-R, a scale for assessment of procedural pain. | At one occasion during the study period (72 hours) when the analgesic treatment has not been changed the last six hours.
  Procedural pain response at a short standardized pain stimulation; as scored by a procedural pain assessment scale (Premature Infant Pain Profile - revised, PIPP-R) in relation to PK. The relation to PK will be analysed with NONMEM statistics.
Pharmacogenetic profile in relation to PK results how PK phenotypes depend on pharmacogenetic (PG) profiles. | One blood sample during the study period of 72 hours
  Whole exome sequencing will be conducted, specific pain related genes investigated and related to PK
Pharmacogenetic profile in relation to PD results | One blood sample during the study period of 72 hours
  Whole exome sequencing will be conducted, specific pain related genes investigated and related to pain response as assessed with scores, serum cortisol and skin conductance.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Norman, MD, Principal Investigator — Region Skane
Locations (2):
- Sweden (2):
  - Skane University Hospital, Lund
  - Marco Bartocci, Stockholm

IPD SHARING:
Plan to Share IPD: No